CLINICAL TRIAL: NCT04963257
Title: A Randomized Controlled Trial of Sertraline Combined With Fluvoxamine in the Treatment of Refractory Obsessive-compulsive Disorder
Brief Title: Sertraline Combined With Fluvoxamine in the Treatment of Refractory Obsessive-compulsive Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-234
Record Dates: First submitted 2019-11-17; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: OCD
Keywords: sertraline; OCD; fluvoxamine
MeSH Terms: interventions — Fluvoxamine; Sertraline; Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sertraline combined with fluvoxamine (Experimental): Sertraline combined with fluvoxamine treatment group: Gradually add the drug to the treatment dose, and monitor the symptom change, scale score, blood drug concentration and other indicators
  Interventions: Drug: sertraline fluvoxamine
- sertraline combined with aripiprazole (Active Comparator): sertraline combined with aripiprazole treatment group:Gradually add the drug to the treatment dose, and monitor the symptom change, scale score, blood drug concentration and other indicators
  Interventions: Drug: sertraline

INTERVENTIONS:
Drug: sertraline fluvoxamine — the initial dose of sertraline was given 50mg/d and the initial dose of fluvoxamine was 50mg/d, and the target dose of sertraline was gradually increased to 200mg/ d and the target dose of fluvoxamine was 200-300mg/d within 2 weeks, and the specific dose adjustment process was determined by the doctors on the basis of patients' conditions
  Other Names: fluvoxamine
  Arms: sertraline combined with fluvoxamine
Drug: sertraline — The initial dose of sertraline was 50mg/d and the initial dose of aripiprazole was 5mg/d. The target dose of sertraline was 200mg/ d and the target dose of aripiprazole was 5-20mg/d within 2 weeks, and the specific dose adjustment process was determined by the doctors on the basis of patients' conditions
  Other Names: aripiprazole
  Arms: sertraline combined with aripiprazole

SUMMARY:
To verify that sertraline combined with fluvoxamine is superior to sertraline combined with aripiprazole

DETAILED DESCRIPTION:
To verify that sertraline combined with fluvoxamine is superior to sertraline combined with aripiprazole, and to observe the indicators of improving patients' cognitive function and adverse drug reactions, so as to provide evidence-based evidence for supplementing the treatment guidelines for obsessive-compulsive disorder

ELIGIBILITY:
Inclusion Criteria:

* The Diagnostic criteria of OCD in the Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-V), as well as the definition of refractory OCD, are as follows: failure to respond to oral treatment with at least two effective doses of antidepressants, including: Fluoxetine (≥20mg/ d), fluvoxamine (≥200mg/d), sertraline (≥150mg/d), and paroxetine (≥ 40mg/d) were all treated for at least 12 weeks. The Yale-Brown compulsive scale (Y-BOCS) score decreased by < 35%.
* The total score of Yale- Brown compulsion scale (Y-BOCS) ≥16 points. (3)age 12 ~ 45 years.

Exclusion Criteria:

* Exclusion of severe organic brain disease;
* Severe physical illness;
* Other mental disorders such as tics, disruptive disorders, eating disorders and autism spectrum disorders;
* Pediatric streptococcal infection causedby autoimmune neuropsychiatric disease (PANDAS);
* Alcohol and drug dependence; Angle-closure glaucoma;
* Suicidal tendencies;
* Previous history of drug allergies related to research;
* Pregnant and lactating women.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Y-BOCS score | 12 weeks
  Treatment effectiveness was defined as a reduction of ≥35% in Y-BOCS score compared to baseline(12 weeks). Treatment recovery: Y-BOCS score below 8 (12 weeks)
Ratio of Y-BOCS score reduction from baseline | 12 weeks
  Treatment effectiveness was defined as a reduction of ≥35% in Y-BOCS score compared to baseline(12 weeks).

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Affiliated Hospital of Zhejiang University Medical College, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes